CLINICAL TRIAL: NCT03648827
Title: Phase 2 Clinical Pharmacology Study to Assess Dystrophin Levels in Subjects With nmDMD Before and After Treatment With Ataluren
Brief Title: A Study to Assess Dystrophin Levels in Participants With Nonsense Mutation Duchenne Muscular Dystrophy (nmDMD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC124-GD-045-DMD; 2019-001767-67 (EudraCT Number)
Record Dates: First submitted 2018-08-24; First posted 2018-08-27 (Actual); Results first posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-02

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — ataluren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ataluren (Experimental): Participants will receive ataluren oral suspension 10 milligrams per kilogram (mg/kg) in the morning, 10 mg/kg at midday, and 20 mg/kg in the evening each day for 40 weeks.
  Interventions: Drug: Ataluren

INTERVENTIONS:
Drug: Ataluren — Ataluren will be administered as per the dose and schedule specified in the arm.
  Other Names: PTC124

SUMMARY:
This study is designed to evaluate the ability of ataluren to increase dystrophin protein levels in muscle cells of participants with nmDMD. The study will evaluate the levels of dystrophin before and after 40 weeks of ataluren therapy using muscle biopsies and 2 validated assay methods, electrochemiluminescence (ECL) and immunohistochemistry.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of signed and dated informed consent/assent document(s) indicating that the participant (and/or his parent/legal guardian) has been informed of all pertinent aspects of the trial.
* Phenotypic evidence of duchenne muscular dystrophy (DMD) based on the onset of characteristic clinical symptoms or signs (for example, proximal muscle weakness, waddling gait, and Gowers' maneuver) and an elevated serum creatine kinase (CK). Medical documentation of phenotypic evidence of DMD needs to be provided upon request by the Sponsor's medical monitor.
* Documentation of the presence of a nonsense point mutation in the dystrophin gene as determined by gene sequencing. Review and approval of documentation by sponsor or designee is required prior to enrollment.
* Willing to undergo muscle biopsy.

Exclusion Criteria:

* Ongoing intravenous (IV) aminoglycoside or IV vancomycin therapy.
* Known contra-indication to muscle biopsy (such as bleeding or clotting disorders).
* Prior or ongoing therapy with ataluren.
* Known hypersensitivity to any of the ingredients or excipients of the study drug (for example, refined polydextrose, polyethylene glycol 3350, poloxamer 407, mannitol 25C, crospovidone XL10, hydroxyethyl cellulose, colloidal silica, magnesium stearate).
* Exposure to another investigational drug within 2 months prior to start of study treatment, or ongoing participation in any interventional clinical trial.
* Requirement for daytime ventilator assistance or any use of invasive mechanical ventilation via tracheostomy. Evening non-invasive mechanical ventilation such as use of bilevel positive airway pressure (Bi-PAP) therapy is allowed.
* Elevated serum creatinine or cystatin C levels at screening.
* Prior or ongoing medical condition (for example, concomitant illness, psychiatric condition, behavioral disorder), medical history, physical findings or laboratory abnormality that, in the investigator's opinion, could adversely affect the safety of the participant, makes it unlikely that the course of treatment or follow-up would be completed, or could impair the assessment of study results.

Ages: 2 Years to 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Bibbiani, MD, Study Director — PTC Therapeutics, Inc.
Locations (9):
- United States (9):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - University of California (UC) Davis Medical Center, Sacramento, California
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University College of Physicians & Surgeons, New York, New York
  - Texas Children's Hospital, Houston, Texas
  - University of Texas Heath Science Center at San Antonio, San Antonio, Texas
  - Children's Hospital of the King's Daughters, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Ataluren: Participants received ataluren oral suspension 10 milligrams per kilogram (mg/kg) in the morning, 10 mg/kg at midday, and 20 mg/kg in the evening each day for 40 weeks.
Period: Overall Study
Arm/Group | Ataluren
Started | 20
Received at Least 1 Dose of Study Drug | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all enrolled participants with a valid assessment of dystrophin level at baseline, as measured by electrochemiluminescence (ECL).
Groups:
- Ataluren: Participants received ataluren oral suspension 10 mg/kg in the morning, 10 mg/kg at midday, and 20 mg/kg in the evening each day for 40 weeks.
Arm/Group | Ataluren
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.8 (1.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 17
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Dystrophin Level at Week 40, as Measured by ECL
Description: The percent change in dystrophin level from baseline in ambulatory nonsense mutation duchenne muscular dystrophy (nmDMD) participants after treatment with ataluren for 40 weeks was analyzed using quantitative assay (ECL).The least square (LS) mean and 90% confidence interval (CI) were analyzed from a mixed-model repeated measures (MMRM) with factors of muscle locations and visits as fixed effects, and participants as a random effect.
Time Frame: Baseline, Week 40
Population: ITT population included all enrolled participants with a valid assessment of dystrophin level at baseline, as measured by ECL.
Measure: Least Squares Mean (90% Confidence Interval); unit: percent change
Arm/Group | Ataluren
Number analyzed (Participants) | 20
percent change | 6.559 [-8.402 to 23.963]

2. Secondary Outcome: Percent Change From Baseline in Dystrophin Level at Week 40, as Determined by Immunohistochemistry (IHC) Membrane Stain Density
Description: The percent change in dystrophin level from baseline in ambulatory nmDMD participants after 40 weeks of ataluren therapy was determined by IHC membrane stain density. The LS mean and 90% CI were analyzed from an MMRM with factors of muscle locations and visits as fixed effects, and participants as a random effect.
Time Frame: Baseline, Week 40
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: percent change
Arm/Group | Ataluren
Number analyzed (Participants) | 20
percent change | 4.914 [-1.642 to 11.906]

ADVERSE EVENTS:
Time Frame: Baseline up to Week 40
Description: Safety Population included all participants who received at least 1 dose of ataluren.
Arm/Group | Ataluren
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 2/20
Other Adverse Events (participants affected / at risk) | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ataluren (N=20)
COVID-19 (Infections and infestations) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ataluren (N=20)
Diarrhoea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 2
Gait inability (General disorders) | 1
Oedema peripheral (General disorders) | 1
Ear infection (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
COVID-19 (Infections and infestations) | 1
Conjunctivitis bacterial (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Pharyngitis streptococcal (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Procedural pain (Injury, poisoning and procedural complications) | 6
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 3
Femur fracture (Injury, poisoning and procedural complications) | 1
Urine output increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Aggression (Psychiatric disorders) | 1
Behaviour disorder (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Miliaria (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results and/or communications prior to public release and can embargo communications regarding trial results for a period that is up to 180 days from the time submitted to the sponsor for review. The sponsor may consult with the PI to require changes to the communication or extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT03648827/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/27/NCT03648827/SAP_001.pdf